CLINICAL TRIAL: NCT03201367
Title: Efficacy and Safety of Rivaroxaban in the Management of Acute Non-neoplastic Portal Vein Thrombosis in HCV Related Compensated Cirrhosis
Brief Title: Efficacy and Safety of Rivaroxaban in Acute Non-neoplastic Portal Vein Thrombosis in HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Shaaban Hanafy, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3779
Record Dates: First submitted 2017-05-26; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Portal Vein Thrombosis
Keywords: Portal vein; thrombosis; acute; rivaroxaban
MeSH Terms: conditions — Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: 40 patients received rivaroxaban
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): acute non-neoplastic PVT, compensated cirrhosis, acute PVT onset within 1 week after initial diagnosis
  - treated with rivaroxaban
  Interventions: Drug: Rivaroxaban
- control group (Placebo Comparator): acute non-neoplastic PVT, compensated cirrhosis, acute PVT onset within 1 week after initial diagnosis receive placebo
  Interventions: Other: symptomatic therapy for ascites, abdominal pain

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 10 mg/12 hour
  Arms: study group
Other: symptomatic therapy for ascites, abdominal pain
  Arms: control group

SUMMARY:
Portal vein thrombosis (PVT) in patients with liver cirrhosis may be due to neoplastic growth or non-neoplastic causes.

* Treating PVT with anticoagulation in liver cirrhosis is difficult to be established but may be of great benefit in acute symptomatic PVT.
* The ultimate goal is complete recanalization of the portal vein without inducing major bleeding, abnormal liver function tests or increased mortality.

DETAILED DESCRIPTION:
Out of 220 patients with chronic HCV who had undergone splenectomy due to hypersplenism in the period extending from May 2014 until August 2016; 36 participants (16.4%) were selected. They were presented with acute PVT. Also, the investigators enrolled 4 patients who were presented with PVT due to portal pyemia complicated infected thrombosed internal piles (n=1), appendicular abscess (n=1), ulcerative colitis (n=2).

Control group It included 30 patients who had acute non-neoplastic PVT with the same inclusion criteria and were given symptomatic therapy for ascites, abdominal pain and followed synchronously with the study group.

Laboratory investigations They included investigation preliminary to splenectomy as liver function tests, coagulation profile, renal function tests, complete blood count, reticulocyte count and bone marrow aspiration. For each patient, Child-Pugh (CTP) and MELD scores were calculated.

Abdominal Ultrasonography (USG) Cirrhotic echo pattern, criteria of portal hypertension, ascites, HCC were excluded Color Doppler Sonography to confirm the diagnosis of PVT. Upper GI Endoscopy All the patients before splenectomy were exposed to upper GI endoscopy to detect the presence and grading of gastro-esophageal varices.

Protocol of therapy Enoxaparin was initiated at a dose of 1mg/kg every 12 hours subcutaneously for 3 days then treatment was continued with rivaroxaban 10mg/12 hr. Rivaroxaban was started 2 hours before the next dose of enoxaparin.

* Follow up every week with a questionnaire about symptoms of bleeding (hematemesis, melena, epistaxis, gum bleeding, vaginal bleeding, subcutaneous bleeding), worsening or improvement of abdominal pain.
* Bedside ultrasonography for detection of thrombus resolution and presence or improvement of ascites every 2 weeks Laboratory follow-up which included serum creatinine, complete blood count, and liver function tests to detect if there any side effects of the therapy every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Acute non-neoplastic portal vein thrombosis
* Compensated cirrhosis (Child class A-B)
* The onset of PVT is within 1 week.

Exclusion Criteria:

* Decompensated liver disease
* Bleeding tendency or recent bleeding event as bleeding peptic ulcer or oesophageal varices
* Neoplastic invasion of the portal vein
* Renal impairment with the creatinine clearance ≤ 30 ml/min
* Pregnancy and breastfeeding
* Hypersensitivity to rivaroxaban
* Concomitant treatment with another anticoagulant
* Concomitant use of clopidogrel.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
complete recanalization of the portal vein | 6 months
  bedside ultrasonography for detection of thrombus resolution

SECONDARY OUTCOMES:
major bleeding | 6 months
  Questionnaire about symptoms of bleeding (hematemesis, melena, epistaxis, gum bleeding, vaginal bleeding, subcutaneous bleeding)
Hepatotoxicity | 6 MONTHS
  liver function tests as AST, ALT (IU/L), total bilirubin (mg/dl)

OTHER OUTCOMES:
short term survival | 1 year
  impact of treating portal vein thrombosis on short term survival

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hanafy AS, Abd-Elsalam S, Dawoud MM. Randomized controlled trial of rivaroxaban versus warfarin in the management of acute non-neoplastic portal vein thrombosis. Vascul Pharmacol. 2019 Feb;113:86-91. doi: 10.1016/j.vph.2018.05.002. Epub 2018 Jun 7. PMID 29886103